CLINICAL TRIAL: NCT07047924
Title: A Prospective, Multi-centre, Single-Arm Clinical Trial of Orthokeratology Lenses (MCOK-01) in Subjects With Myopia and Myopic Astigmatism
Brief Title: A Clinical Trial Assessing the Safety and Effectiveness of Orthokeratology Lenses in Patients With Myopia and Myopic Astigmatism
Acronym: SEMOA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Menicon Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCOK-3-AUS
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Myopia; Myopic Astigmatism
Keywords: Myopia; Myopic Astigmatism; Orthokeratology Lenses; Orthokeratology
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- Investigational (Experimental): All participants will be enrolled in the Investigational arm, and treated with the investigational product.
  Interventions: Device: MCOK-01

INTERVENTIONS:
Device: MCOK-01 — The investigational device is a Rigid Gas Permeable contact lenses for orthokeratology. MCOK-01 applied the reverse geometry design and adopted the lens material which possesses the highest oxygen permeability among all the materials for orthokeratology lens.

SUMMARY:
This is a prospective, multi-centre, single-arm clinical trial to evaluate the effectiveness and safety of MCOK-01 lenses in patients with myopia and myopic astigmatism who need dioptric correction.

A maximum number of 220 participants are planned to be enrolled , with a minimum of 150 planned to complete the trial (30% dropout). All participants will be enrolled in Australia.

Enrolled participants will wear the lenses every night for up to 12 months, removing them upon waking. 8 follow up visits will be completed during treatment, after: 1 day, 1 week, 2 weeks, 1 month, 3 months, 6 months, 9 months and 12 months of wearing the lenses.

ELIGIBILITY:
Inclusion Criteria:

1. Participant diagnosed with myopia and myopic astigmatism, documented by an eye care practitioner.
2. Participant is between 6-40 years old inclusive.
3. Participant is not motivated to wear glasses in daily life.
4. Participants are of Caucasian ethnicity (must be >50% of study population) or other non-east Asian ethnic groups (Indian, Sri-Lankan, Pakistani, etc). Neither parent of participant can be east-asian.
5. Provision of written informed consent.
6. Participants understand and agree to all requirements of the clinical trial; visit schedule, investigator guidance, follow-lens instructions, etc

Exclusion Criteria:

1. Best corrected distance vision acuity of less than 0.8 with spectacles.
2. Subjective refraction test shows spherical power greater than -6.00D,less than -0.50D or astigmatism greater than 1.5D.
3. Participants of East-Asian ethnicity (Chinese, Japanese, Korean, etc).
4. Participants requiring treatment for eye disease other than refractive error (excluding those receiving artificial tears eye drops due to the wearing of corneal contact lenses).
5. Medical history of intraocular surgery that may affect the effect of wearing the lens for this clinical trial (those with corneal transplantation, Retinal detachment, etc)..
6. Medical history of refractive corneal surgery.
7. Slit lamp findings that are more serious than grade 1
8. Participants requiring lens parameters outside of the scope of lens for this clinical trial.
9. Known eye allergies or conditions that are contraindicated, including sensitivity to any lens care maintenance or packaging solution additives being used in this study
10. Corneal abnormalities including keratoconus, corneal dystrophy and/or previous history of ocular herpes infections.
11. Currently using Atropine, or have used Atropine eye drops 14 days prior to enrolment.
12. For female participants, pregnancy, planned pregnancy during the trial or breastfeeding (pregnancy status provided by verbal confirmation).
13. Participation in other clinical trials or participation within the past 30 days.
14. Use of orthokeratology lenses within the prior 90 days, extended wear, rigid gas permeable corneal and scleral lenses within the prior 30 days, daily disposable and daily wear within the prior 15 days.
15. Mental incapacity.
16. Other Participants deemed not suitable for the trial at the investigator's discretion

Ages: 6 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Lines of improvement of monocular uncorrected distance visual acuity | 12-months following enrolment
  Reading of a logMAR chart. Each line difference represents 0.1 logMAR acuity. The improvement in acuity is represented by a numerical reduction in the logMAR value.
Proportion of eyes achieved uncorrected distance visual acuity of ≤0.30 logMAR, ≤0.20 logMAR, ≤0.10 logMAR, and ≤0.00 logMAR | 1 month, 3 months, 6 months, 9 months, and 12 months following enrolment
  Measured using a logMAR chart. Each line difference represents 0.1 logMAR acuity. The improvement in acuity is represented by a numerical reduction in the logMAR value.
A level of attempted versus achieved reduction in manifest refractive error | 12 months following enrolment
  Using a Phoropter/Refractor. Proportion of eyes with manifest sphere within ±0.50 D, ±1.00 D, and ±2.00 D of the target (plano)
Number and rates (by type of event and relation to device) of serious and significant adverse events | Any time within the 12-months enrolment window
  Adverse events will be self-reported by participants to investigative team
Number and rates (by type of event) of all types of adverse events that were not classified as serious or significant adverse events. | Any time within the 12-months enrolment window
  Adverse events will be self-reported by participants to investigative team
Number of slit lamp results above grade 2 | 1 day, 1 week, 2 weeks, 1 month, 3 months, 6 months, 9 months, and 12 months following enrolment
  Assessed using a slit lamp
Number and rate of cases of loss of; monocular best spectacle corrected visual acuity (BSCVA) of 2 or more lines (≥ 0.2 logMar), and 1 or more lines (≥ 0.1 logMar). | 1 day, 1 week, 2 weeks, 1 month, 3 months, 6 months, 9 months, and 12 months following enrolment
  Assessed with a logMAR chart

SECONDARY OUTCOMES:
Improvement of monocular uncorrected distance visual acuity | 1 month, 3 months, 6 months, 9 months, and 12 months following enrolment
  Assessed with a logMAR chart. Endpoint will be measured by a set of descriptive statistics.
Change in best corrected spectacle visual acuity | 1 day, 1 week, 2 weeks, 1 month, 3 months, 6 months, 9 months, and 12 months following enrolment
  Assessed using a logMAR chart
Changes in manifest sphere | 1 month, 3 months, 6 months, 9 months, and 12 months following enrolment
  Measured with a subjective refraction test
A level of attempted versus achieved reduction in manifest refractive error | 1 month, 3 months, 6 months, 9 months, and 12 months following enrolment
  Measured with a subjective refraction test. Proportion of eyes with manifest sphere within ±0.50 D, ±1.00 D, and ±2.00 D of the target (plano)
Corneal topography changes | 12 months following enrolment
  Measured with a corneal topographer
Change in absolute corneal astigmatism | 12 months following enrolment
  Measured with a corneal topographer
Number of discontinued participants and the reasons for discontinuation | Any time within the 12-months enrolment window
  Ongoing participation rates will be continuously monitored
Number and rates of average wear time per day | 1 day, 1 week, 2 weeks, 1 month, 3 months, 6 months, 9 months, and 12 months following enrolment
  Patient reported at scheduled study visits
Increase in corneal or refractive astigmatism of 2D or more and 1D or more post-treatment | 12 months following enrolment
  Measured with a subjective refraction test
Signs/symptoms and complications from subjective questionnaires | 1 month, 6 months, and 12 months following enrolment
  Assessed by the subjective questionnaires completed by participants
Descriptive statistics of intraocular pressure (IOP) and for percent change from baseline | 6 months and 12 months following enrolment
  Measured using a tonometer
Descriptive statistics of specular microscopy measurements | 12 months following enrolment
  Measured using a specular microscope. Specific parameters include Endothelial Cell Morphology (Cell density (cells/mm2), Polymegethism (CV) and Pleomorphism (percentage of hexagonal cells))
Descriptive statistics of central corneal thickness | 6 months, and 12 months following enrolment
  Measured using a specular microscope.
Frequency and reasons for lens replacement | Any time within the 12-months enrolment window
  Patient reported at scheduled study visits
Damage or scratches on the lenses | 1 day, 1 week, 2 weeks, 1 month, 3 months, 6 months, 9 months, and 12 months following enrolment
Stability in manifest refractive error | 1 month and 3 months following enrolment
  Measured with a subjective refraction test. Proportion of eyes with manifest sphere change within ±0.50 D between 1-month and 3-month visit.
Stability in unaided visual acuity | 1 month and 3 months following enrolment
  Measured using a logMAR chart. Proportion of eyes with unaided visual acuity change within 1 line (0.1 logMAR) between 1-month and 3-month visit.

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - Eyecare Kids, Hillsdale, New South Wales
  - UNSW School of Optometry and Vision Science, Sydney, New South Wales
  - Queensland University of Technology Optometry and Vision Science, Kelvin Grove, Queensland
  - The University of Melbourne Department of Optometry and Vision Sciences, Carlton, Victoria

IPD SHARING:
Plan to Share IPD: No